CLINICAL TRIAL: NCT05673993
Title: A Phase Ⅲ, Multi-center, Randomized, Placebo-controlled, Study to Evaluate the Efficacy and Safety of Subcutaneous Telitacicept in Subjects With Active Primary Sjogren's Syndrome
Brief Title: A Study to Evaluate the Efficacy and Safety of Telitacicept in Subjects With Active Primary Sjogren's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18C022
Record Dates: First submitted 2022-12-29; First posted 2023-01-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: Primary Sjogren's Syndrome
Keywords: primary Sjogren's Syndrome; pSS; RC18
MeSH Terms: interventions — telitacicept; RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telitacicept 80 mg (Experimental): Subjects will be given subcutaneous Telitacicept 80 mg once a week for 48 weeks.
  Interventions: Biological: Telitacicept 80 mg
- Telitacicept 160 mg (Experimental): Subjects will be given subcutaneous Telitacicept 160 mg once a week for 48 weeks.
  Interventions: Biological: Telitacicept 160 mg
- Placebo (Placebo Comparator): Subjects will be given subcutaneous placebo once a week for 24-48 weeks. Subjects who are randomized to the placebo group are allowed to be transferred to either Telitacicept 80 mg or Telitacicept 160 mg after Week 24 by the investigator. Subjects and investigators are blinded throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept 80 mg — Telitacicept 80 mg subcutaneously once a week.
  Other Names: RC 18 80 mg
  Arms: Telitacicept 80 mg
Biological: Telitacicept 160 mg — Telitacicept 160 mg subcutaneously once a week.
  Other Names: RC 18 160 mg
  Arms: Telitacicept 160 mg
Drug: Placebo — Subjects will be given subcutaneous placebo once a week.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of subcutaneous Telitacicept versus placebo in subjects with active primary Sjogren's Syndrome.

DETAILED DESCRIPTION:
This is a phase Ⅲ, multi-center, randomized, double-blind, placebo-controlled study. Subjects with active primary Sjogren's Syndrome (pSS) will be randomized to receive subcutaneous Telitacicept 80 mg, Telitacicept 160 mg or placebo weekly for a total of 48 weeks. Subjects are allowed to be transferred to another group after Week 24 by the investigator so that those randomized to the placebo group are able to receive either Telitacicept 80 mg or Telitacicept 160 mg afterwards. Subjects who are randomized to Telitacicept 80 mg and Telitacicept 160 mg groups will remain in the previous treatment group even if the investigator chooses to transfer them. Subjects and investigators are blinded throughout the study.

ELIGIBILITY:
Main Inclusion Criteria:

1. Written informed consent provided.
2. Males and females, 18-70 years of age.
3. Fulfilled the classification criteria of pSS according to ACR/EULAR (2016).
4. Anti-SSA antibody tested positive at screening.
5. ESSDAI score ≥ 5 at screening.

Main Exclusion Criteria:

1. Secondary Sjogren's syndrome.
2. Severe organ involvement related to pSS in the opinion of the investigator, including but not limited to a) severe vasculitis (not cutaneous vasculitis) affecting the kidney, gastrointestinal system, cardiac, pulmonary or central nervous system (CNS); b) active CNS or peripheral nervous system involvement requiring high dose corticosteroids; c) severe kidney involvement, e.g. GFR < 60 ml/min, serum creatinine > 2 mg/dL, or proteinuria > 3g/d; d) severe pulmonary involvement, e.g. shortness of breath at rest, FVC < 60% or DLCO < 40%; e) muscle diseases requiring high dose corticosteroids; f) lymphoma.
3. Received sodium hyaluronate eye drops, artificial tears or artificial saliva within 7 days prior to screening.
4. Received live vaccine within 28 days prior to randomization.
5. Active hepatitis or history of severe liver diseases.
6. HIV positive.
7. Patients with malignant tumors.
8. Received investigational pharmaceutical within 28 days or 5 half-lives prior to randomization, whichever is longer.
9. Nursing or pregnant female, or male or female who prepared for parenthood during the study.
10. Any condition that, in the opinion of the investigator, makes it unsuitable for the subject to participate, e.g., poorly controlled high blood pressure, diabetes, heart failure or mental illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ESSDAI score | Week 24
  The EULAR Sjogren's syndrome (SS) disease activity index (ESSDAI) is a systemic disease activity index that was designed to measure disease activity in patients with primary SS. It includes 12 domains (ie, organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular, constitutional, lymphadenopathic, biological). Each domain is divided into 3-4 levels of activity (no, low, moderate, high). Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity). A higher score indicates worsening of the disease.

SECONDARY OUTCOMES:
Change from baseline in ESSDAI score | Week 48
  The EULAR Sjogren's syndrome (SS) disease activity index (ESSDAI) is a systemic disease activity index that was designed to measure disease activity in patients with primary SS. It includes 12 domains (ie, organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular, constitutional, lymphadenopathic, biological). Each domain is divided into 3-4 levels of activity (no, low, moderate, high). Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity). A higher score indicates worsening of the disease.
Percentage of subjects with ESSDAI score decreased from baseline by at least 3 points | Week 24 & Week 48
  The EULAR Sjogren's syndrome (SS) disease activity index (ESSDAI) is a systemic disease activity index that was designed to measure disease activity in patients with primary SS. It includes 12 domains (ie, organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular, constitutional, lymphadenopathic, biological). Each domain is divided into 3-4 levels of activity (no, low, moderate, high). Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity). A higher score indicates worsening of the disease
Percentage of subjects with ESSDAI score < 5 | Week 24 & Week 48
  The EULAR Sjogren's syndrome (SS) disease activity index (ESSDAI) is a systemic disease activity index that was designed to measure disease activity in patients with primary SS. It includes 12 domains (ie, organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular, constitutional, lymphadenopathic, biological). Each domain is divided into 3-4 levels of activity (no, low, moderate, high). Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity). A higher score indicates worsening of the disease.
Percentage of subjects with ESSPRI score decreased from baseline by at least 1 point or 15% | Week 24 & Week 48
  The EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) is a patient-reported, subjective symptom index for primary Sjögren's syndrome. It consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains.
Change from baseline in MFI-20 | Week 24 & Week 48
  The multidimensional fatigue inventory (MFI-20) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue. Each question is scored from one to five and each dimension consists of five questions. The dimensional score consequently ranges from 4 to 20 (a higher score indicates more fatigue).
Incidence of AEs, SAEs | Up to Week 48
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death; is life-threatening experience; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/ birth defect; or any other important medical event that may not be immediately life-threatening or result in death or hospitalization but may require intervention to prevent one of the other serious outcomes listed in the definition above.

CONTACTS AND LOCATIONS:
Locations (78):
- China (78):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - South China Hospital of Shenzhen University, Shenzhen, Guangdong
  - Zhongshan Hospital of Traditional Chinese Medicine, Zhongshan, Guangdong
  - Guilin People's Hospital, Guilin, Guangxi
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Hebei PetroChina Central Hospital, Langfang, Hebei
  - The Second Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First People's Hospital of Changde, Changde, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Chenzhou, Chenzhou, Hunan
  - The Second People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - Yanbian University Hospital (Yanbian Hospital), Yanji, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Jining No 1 People's Hospital, Jining, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Yantaishan Hospital, Yantai, Shandong
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hopital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Huzhou Third Municipal Hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The Second Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Ningbo Medical Center (Lihuili Hospital), Ningbo, Zhejiang
  - The First People's Hospital of Wenling, Wenling, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The People's Hospital of Wenzhou, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided